CLINICAL TRIAL: NCT05962814
Title: EarGenie: Assessment of a Minimum Viable Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Bionics Institute of Australia (Other)
Responsible Party: Principal Investigator, Colette McKay, Leader, Translational Hearing Research and Principal Scientist, The Bionics Institute of Australia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 98058
Record Dates: First submitted 2023-07-10; First posted 2023-07-27 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Hearing Impaired Children
Keywords: fNIRS; Early intervention

STUDY DESIGN:
Intervention Model Description: A single group of infants without hearing impairment will be recruited so that safety and preliminary efficacy can be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fNIRS (Experimental): Infants who have a test completed with EarGenie MVP in a single test session
  Interventions: Device: EarGenie MVP test

INTERVENTIONS:
Device: EarGenie MVP test — The EarGenie test consists of placing the EarGenie headgear on the infant and running the fNIRS tests via the user interface. Blocks of speech sounds are presented to the infant via earphones or via speaker, and the EarGenie MVP measures changes in the blood oxygenation. Automatic analyses are run to determine whether the infant heard the sounds or discriminated between them. The infant will be in a natural sleep when the fNIRS test is run. Prior to the test, standard audiometric procedures (otoscopy and tympanometry) will confirm normal middle ear function.

SUMMARY:
The goal of this clinical trial is to evaluate safety and preliminary efficacy of a novel device (EarGenie MVP) to assess hearing function in infants, using a small number of infants with normal hearing. The main questions it aims to answer are:

* Is our device safe?
* Does the device provide preliminary results consistent with previous results from a commercial functional Near Infrared Spectroscopy (fNIRS) research device?

Participants will attend one test session and have their hearing assessed with the EarGenie MVP device.

DETAILED DESCRIPTION:
This is a first-in-human study to evaluate safety and preliminary efficacy of our prototype hearing assessment system (EarGenie MVP). EarGenie MVP uses fNIRS technology to assess an infant's brain response to hearing speech sounds, or discriminating between different speech sounds. It includes software to automatically run analysis in real time, and has a user interface allowing clinicians to operate the tests and receive result reports. The test methods and analysis software have been developed using our commercial fNIRS research system, but the EarGenie MVP has been designed for easy use in paediatric audiology clinics.

10 infants with normal hearing will be recruited for the study, and undergo one test session each with the EarGenie MVP. Safety data will be documented and the results of the tests examined to see if they are consistent with the results expected from our experience using the commercial device in 36 infants with normal hearing.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 1 and 24 months at the time of fNIRS testing.
* Has no known hearing loss
* Has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.

Exclusion Criteria:

* There are no exclusion criteria other than not meeting the inclusion criteria.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colette M McKay, PhD, Principal Investigator — The Bionics Institute of Australia
Locations (1):
- Bionics Institute, East Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 Participants were recruited via word of mouth between August 2023 and February 2024.
Pre-assignment Details: One infant was found to have middle ear disfunction on the tympanometry test, and so was excluded from the study and did not complete an fNIRS test
Period: Overall Study
Arm/Group | fNIRS
Started | 11
Completed | 10
Not Completed | 1
Not completed — failed eligibility | 1

BASELINE CHARACTERISTICS:
Arm/Group | fNIRS
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants] — Age of infants noted via birth dates
  Participants
    1-24 months | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 10

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Significant fNIRS Detection and Discrimination Responses
Description: Evidence of device feasibility will be obtained by comparing the test results obtained using EarGenie MVP to our existing test results for a larger number of infants obtained with a commercial device NIRx (McKay et al. 2023. "A Reliable, Accurate, and Clinic-friendly Objective Test of Speech Sound Detection and Discrimination in Sleeping Infants." PsyArXiv. June 20. doi:10.31234/osf.io/fbwcm).
  For each infant, the presence of a significant response is determined by the incorporated automatic analysis software, and further visually supported for the tester by checking that the shape of the response waveform is consistent with those found in the previous data set. We will consider the feasibility as confirmed if not more than 1(/10) infants (or 10%) have an absent detection response at 65 dB SPL, and not more than 3 (/10) babies (or 30%) show an absent discrimination response for "Ba" versus "Ga".
Time Frame: Each infant has one test session, lasting up to to hours. Outcome measures are determined after the last infant has been tested.
Measure: Count of Participants; unit: Participants
Arm/Group | fNIRS
Number analyzed (Participants) | 10
Participants
  significant detection response to BA at 65 dB SPL: with | 4
  significant detection response to BA at 65 dB SPL: without | 6
  significant discrimination response to BA/GA contrast: with | 1
  significant discrimination response to BA/GA contrast: without | 9
  Response morphologies consitent with morphologies of research device: with | 10
  Response morphologies consitent with morphologies of research device: without | 0

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Safety assessment will be undertaken as follows. Any adverse event (as defined using standard definitions) will be documented in each infant's case report, and reported using standard required procedures. Each infant's case report will also include details of any minor non-reportable occurrences only relevant to comfort of use such as discomfort signs in the infant, or any temporary visual skin marks left by the headgear after the test.
  If any major adverse effect occurs, the trial will be stopped until the such time as the issue is resolved.
Time Frame: Adverse effects are noted during, and for 24 hours following the single test session of the infant. Incidence of events is calculated after the last infant is tested.
Measure: Count of Participants; unit: Participants
Arm/Group | fNIRS
Number analyzed (Participants) | 10
Participants
  Adverse events: with | 0
  Adverse events: without | 10
  no impression marks on skin, or impression marks that resolved within 3 hours: with | 10
  no impression marks on skin, or impression marks that resolved within 3 hours: without | 0
  signs of distress during test such as crying: with | 0
  signs of distress during test such as crying: without | 10

ADVERSE EVENTS:
Time Frame: Data were collected over the duration of the trial, and for each infant during the test and the 24 hours post the test
Arm/Group | fNIRS
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT05962814/Prot_SAP_000.pdf